CLINICAL TRIAL: NCT02049905
Title: A Multicenter, Randomized, Open-Label Phase 3 Study to Investigate the Efficacy and Safety of Aldoxorubicin Compared to Investigator's Choice in Subjects With Metastatic, Locally Advanced, or Unresectable Soft Tissue Sarcomas Who Either Relapsed or Were Refractory to Prior Non-Adjuvant Chemotherapy
Brief Title: Phase 3 Study to Treat Patients With Soft Tissue Sarcomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P3-STS-01
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2017-06

CONDITIONS: Metastatic, Locally Advanced or Unresectable Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; unresectable; metastatic; locally advanced; sarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma | interventions — DOXO-EMCH; pazopanib; Gemcitabine; Docetaxel; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aldoxorubicin (Experimental): Aldoxorubicin is administered at 350 mg/m2 (260 mg/m2 doxorubicin equivalent) intravenously on Day 1 every 21-day cycles until tumor progression or unacceptable toxicity occurs.
  Interventions: Drug: Aldoxorubicin
- Investigator's Choice of Treatment (Active Comparator): These treatments include:
  1. Dacarbazine administered at 1000 mg/m2 by intravenous infusion (IVI), over 90±15 minutes on Day 1 every 21 days until tumor progression or unacceptable toxicity occurs;
  2. Pazopanib, 800 mg orally each day until tumor progression or unacceptable toxicity occurs;
  3. Gemcitabine, 900 mg/m2 by IVI over 90 minutes on Days 1 and 8, plus docetaxel, 100 mg/m2 by IVI over 1 hour on Day 8 of a 28 day cycle until tumor progression or unacceptable toxicity occurs;
  4. Doxorubicin, 75 mg/m2 by IVI over 5 to 30 minutes every 21 days for a maximum cumulative dose of 550 mg/m2 or unacceptable toxicity occurs; or
  5. Ifosfamide 2.0 g/m2 administered over 2 to 4 hours on Days 1-4 of a 21 day cycle + mesna per standard site administration regimen until tumor progression or unacceptable toxicity occurs.
  Interventions: Drug: Investigator's Choice Treatment (Darcabazine, Pazopanib, Gemcitabine + Docetaxel, Doxorubicin, Ifosfamide)

INTERVENTIONS:
Drug: Aldoxorubicin
  Other Names: INNO-206
  Arms: Aldoxorubicin
Drug: Investigator's Choice Treatment (Darcabazine, Pazopanib, Gemcitabine + Docetaxel, Doxorubicin, Ifosfamide)
  Other Names: Darcabazine; Pazopanib; Gemcitabine + Docetaxel; Doxorubicin; Ifosfamide
  Arms: Investigator's Choice of Treatment

SUMMARY:
The purpose of this study is to determine the efficacy and safety of aldoxorubicin in subjects with metastatic, locally advanced, or unresectable soft tissue sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent prior to any study related activities.
2. Age ≥15 years (US only), and 18-80 (rest of world (ROW)), male or female.
3. Histological confirmation of intermediate or high grade soft-tissue sarcoma. Tissue must be sent to a central pathology lab for review but will not preclude entry onto the study. Final assignment of tumor grade and histology will be based on the designation provided by the central pathology review.
4. An adequate tumor specimen obtained by either excisional biopsy, incisional biopsy or core needle biopsy must be sent to the central pathology lab for evaluation. The material must measure at least 0.8 × 0.1 cm in size or contain at least 50 tumor cells.
5. Locally advanced, unresectable, and/or metastatic soft-tissue sarcoma of intermediate or high grade with evidence of disease progression by either computed tomography (CT) or magnetic resonance imaging (MRI) scan, or clinical judgment on or after the last cancer therapy within 6 months prior to randomization.
6. Relapsed or refractory (lack of response) to ≥1 course of systemic therapy regimen(s), excluding adjuvant or neoadjuvant chemotherapy, and is incurable by either surgery or radiation.
7. Capable of providing informed consent and complying with trial procedures.
8. ECOG PS 0-2.
9. Life expectancy >12 weeks.
10. Measurable tumor lesions according to RECIST 1.1 criteria.[50]
11. Women must not be able to become pregnant (e.g., post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. (Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.)
12. Males and their female partner(s) of child-bearing potential must use 2 forms of effective contraception (see Inclusion 11 plus condom or vasectomy for males) from the last menstrual period of the female partner during the study treatment and agree to continue use for 6 months after the final dose of study treatment.
13. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
14. Accessibility to the site that optimizes the subject's ability to keep all study-related appointments.

Exclusion Criteria:

1. Prior exposure to >375 mg/m2 of doxorubicin or liposomal doxorubicin.
2. Palliative surgery and/or radiation treatment within 30 days prior to date of randomization.
3. Exposure to any investigational agent within 30 days of date of randomization.
4. Exposure to any systemic chemotherapy within 30 days of date of randomization.
5. An inadequate tumor specimen as defined by the central pathologist.
6. Current evidence/diagnosis of alveolar soft part sarcoma, extraskeletal myxoid chondrosarcoma, rhabdomyosarcoma, osteosarcoma, gastrointestinal stromal tumor (GIST), dermatofibrosarcoma (unless transformed to fibrosarcoma), Ewing's sarcoma, Kaposi's sarcoma, mixed mesodermal tumor, clear cell sarcomas.
7. Evidence of central nervous system (CNS) metastasis who have not received prior definitive therapy for their lesions.
8. History of other malignancies except cured basal cell carcinoma, cutaneous squamous cell carcinoma, melanoma in situ, superficial bladder cancer or carcinoma in situ of the cervix unless documented free of cancer for ≥5 years.
9. Laboratory values: Screening serum creatinine >1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) >3×ULN or >5×ULN if liver metastases are present, total bilirubin >2×ULN, absolute neutrophil count (ANC) <1,500/mm3, platelet concentration <100,000/mm3, hemoglobin <9g/dL.
10. Clinically evident congestive heart failure (CHF) > class II of the New York Heart Association (NYHA) guidelines.
11. Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
12. Baseline QTc >470 msec and/or previous history of QT prolongation while taking other medications.
13. Concomitant use of medications associated with a high incidence of QT prolongation is not allowed.
14. History or signs of active coronary artery disease with or without angina pectoris within the last 6 months.
15. Serious myocardial dysfunction defined by ECHO as absolute left ventricular ejection fraction (LVEF) below the institution's lower limit of predicted normal.
16. Known history of HIV infection.
17. Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals. The Medical Monitor should be contacted for any uncertainties.
18. Major surgery within 30 days prior to date of randomization.
19. Current or past substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
20. Any condition that is unstable and could jeopardize the subject's participation in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, PC, Phoenix, Arizona
  - The University of Arizona, Tucson, Arizona
  - City of Hope Medical Group, Duarte, California
  - Samuel Oschin Cancer Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - U of CO Health Sciences Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Oncology Specialists, SC, Niles, Illinois
  - Kansas City Cancer Center, Overland Park, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Center for Health and Healing, Portland, Oregon
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - U of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Fletcher Allen Health Care, Burlington, Vermont
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Center, Hamilton, Ontario
  - McGill University, Montreal, Quebec
- Instituto Clinico Oncologica del Sur (ICOS), Temuco, Región de la Araucanía, Chile
- Herlev Hospital, Herlev, Denmark
- France (6):
  - Institut Bergonie, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre Georges Francois Leclerc, Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Regional et Universitaire - Hospital Bretonneau, Tours, Centre-Val de Loire
  - Hopital Rene Huguenin - Institut Curie, Saint-Cloud, Île-de-France Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Magyar Honvedseg Egeszsegugyi Kozpont, Budapest, Hungary
- Israel (4):
  - Rambam Medical Center, Haifa
  - Sharet Institute of Oncology Hadassah Ein Karem Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Azienda Ospedaliero-Universitaria di Bologna-Policlinico S Orsola-Malpighi, Bologna
  - IRCCS Instituto Ortopedico Rizzoli, Bologna
  - Istituto Europeo di Oncologia Milano, Milan
  - Istituto Oncologico Veneto, Padua
- Leiden Universitair Medisch Centrum, Leiden, South Holland, Netherlands
- Instytut im.Marii Sklodowskiej-Curie, Warsaw, Poland
- Russia (3):
  - State Institution "Blokhin Cancer Research Centre RAMS", Moscow
  - City Oncology Hospital #2, Moscow
  - Republican Clinical Oncologic Dispensary of Ministry of Health Republic Tatarstan, Tatarstan
- Spain (10):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Inst Catala D'Oncologia, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Hospital de Madrid Norte-San Chinarro, Madrid
  - Hospital San Carlos Madrid, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- See also: Related Info — https://doi.org/10.1093/annonc/mdu354.50
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30936721/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30873850/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29869517/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28846045/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=rubicin%3A+a+tumor-targeted+doxorubicin+conjugate+for+relapsed+or+refractory+soft+tissue+sarcomas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 433 subjects were randomized in the intent to treat population, whereas 420 subjects were in the safety population.
  13 subjects were discontinued prior to treatment start.
Groups:
- Aldoxorubicin: Aldoxorubicin is administered at 350 mg/m2 (260 mg/m2 doxorubicin equivalent) intravenously on Day 1 every 21-day cycles until tumor progression or unacceptable toxicity occurs.
  Aldoxorubicin
- Investigator's Choice of Treatment: These treatments include:
  1. Dacarbazine administered at 1000 mg/m2 by intravenous infusion (IVI), over 90±15 minutes on Day 1 every 21 days until tumor progression or unacceptable toxicity occurs;
  2. Pazopanib, 800 mg orally each day until tumor progression or unacceptable toxicity occurs;
  3. Gemcitabine, 900 mg/m2 by IVI over 90 minutes on Days 1 and 8, plus docetaxel, 100 mg/m2 by IVI over 1 hour on Day 8 of a 28 day cycle until tumor progression or unacceptable toxicity occurs;
  4. Doxorubicin, 75 mg/m2 by IVI over 5 to 30 minutes every 21 days for a maximum cumulative dose of 550 mg/m2 or unacceptable toxicity occurs; or
  5. Ifosfamide 2.0 g/m2 administered over 2 to 4 hours on Days 1-4 of a 21 day cycle + mesna per standard site administration regimen until tumor progression or unacceptable toxicity occurs.
  Investigator's Choice Treatment (Darcabazine, Pazopanib, Gemcitabine + Docetaxel, Doxorubicin, Ifosfamide)
Period: Overall Study
Arm/Group | Aldoxorubicin | Investigator's Choice of Treatment
Started | 218 | 215
Safety Population | 213 | 207
Completed (Completed defined as receiving at least one dose of study drug.) | 213 | 207
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Population: 5 patients were randomized, but not treated on Aldoxorubicin arm. 8 patients were randomized, but not treated on Investigator's Choice of Treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aldoxorubicin | Investigator's Choice of Treatment | Total
Number analyzed (Participants) | 218 | 215 | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (11.68) | 57.0 (12.59) | 56.8 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 128 | 251
  Male | 95 | 87 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 20 | 45
  Not Hispanic or Latino | 178 | 181 | 359
  Unknown or Not Reported | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 13 | 8 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 18 | 23
  White | 174 | 174 | 348
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 24 | 14 | 38
Subjects with Metastatic, Locally Advanced, or Unresectable Soft Tissue Sarcomas Who Either Relapsed [Count of Participants; unit: Participants] | 218 | 215 | 433

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to first documentation of objective tumor progression, according to RECIST 1.1 Criteria, or to death due to any cause in the absence of previous documentation of objective tumor progression. For subjects without documentation of objective tumor progression, who started other anti-tumor treatment, or lost to follow up/withdrew consent prior to confirmed progression, PFS is censored at the date of the last tumor assessment.
  PFS is defined as the interval from the date of randomization to the earliest date of documented evidence of recurrent or progressive disease, or the date of death due to any cause, whichever occurs first.
  PD is defined as: 20% increase in the sum of the longest diameter of target lesions from the smallest sum of the longest diameter recorded since the treatment started; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 new lesion is also considered PD.
Time Frame: 24 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Aldoxorubicin: Aldoxorubicin is administered at 350 mg/m^2 (260 mg/m^2 doxorubicin equivalent) intravenously on Day 1 every 21-day cycles until tumor progression or unacceptable toxicity occurs.
Arm/Group | Aldoxorubicin | Investigator's Choice of Treatment
Number analyzed (Participants) | 218 | 215
Months | 4.04 [2.79 to 4.83] | 2.96 [2.63 to 4.17]

ADVERSE EVENTS:
Time Frame: All AEs that occurred after any administration of the study medication were to be followed until the event resolves, until the subject began alternative treatment, or until 30 days after the last dose of study medication. The SAE reporting period ended if the subject began an alternative therapy or 30 days after the last administration of study drug, up to 640 days.
Groups:
- Aldoxorubicin: Aldoxorubicin is administered at 350 mg/m^2 (260 mg/m^2 doxorubicin equivalent) intravenously on Day 1 every 21-day cycles until tumor progression or unacceptable toxicity occurs.
  Aldoxorubicin
Arm/Group | Aldoxorubicin | Investigator's Choice of Treatment
All-Cause Mortality (participants affected / at risk) | 148/213 | 131/207
Serious Adverse Events (participants affected / at risk) | 91/213 | 68/207
Other Adverse Events (participants affected / at risk) | 209/213 | 203/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldoxorubicin (N=213) | Investigator's Choice of Treatment (N=207)
Febrile neutropenia (Blood and lymphatic system disorders) | 30 | 6
Neutropenia (Blood and lymphatic system disorders) | 11 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Sepsis (Infections and infestations) | 8 | 4
Pneumonia (Infections and infestations) | 3 | 5
Cellulitis (Infections and infestations) | 1 | 4
Bacteraemia (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 2
Small intestine obstruction (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 5 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Malaena (Gastrointestinal disorders) | 1 | 0
Rectal heamorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 5
Asthenia (General disorders) | 2 | 0
Death (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Hypothermia (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Cervial cord compression (Nervous system disorders) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 2
Capillary leak syndrome (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Platelet count decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 4
Mental status change (Psychiatric disorders) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Device occlusion (Product Issues) | 1 | 0
Thrombosis in device (Product Issues) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aldoxorubicin (N=213) | Investigator's Choice of Treatment (N=207)
Nausea (Gastrointestinal disorders) | 108 | 91
Stomatitis (Gastrointestinal disorders) | 114 | 31
Diarrhoea (Gastrointestinal disorders) | 48 | 62
Vomiting (Gastrointestinal disorders) | 60 | 44
Constipation (Gastrointestinal disorders) | 63 | 33
Abdominal Pain (Gastrointestinal disorders) | 32 | 37
Abdominal Pain Upper (Gastrointestinal disorders) | 11 | 10
Dyspepsia (Gastrointestinal disorders) | 8 | 10
Gastroesophageal reflux disease (Gastrointestinal disorders) | 12 | 6
Oral pain (Gastrointestinal disorders) | 12 | 6
Fatigue (General disorders) | 96 | 79
Pyrexia (General disorders) | 34 | 35
Asthenia (General disorders) | 26 | 27
Oedema pheripheral (General disorders) | 22 | 29
Pain (General disorders) | 11 | 11
Anaemia (Blood and lymphatic system disorders) | 96 | 62
Neutropenia (Blood and lymphatic system disorders) | 63 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 29 | 30
Febrile Neutropenia (Blood and lymphatic system disorders) | 32 | 9
Leukopenia (Blood and lymphatic system disorders) | 19 | 10
Decreased Appetite (Metabolism and nutrition disorders) | 60 | 36
Hypokalaemia (Metabolism and nutrition disorders) | 32 | 23
Dehydration (Metabolism and nutrition disorders) | 17 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 16 | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 26
Dyspnoea (Reproductive system and breast disorders) | 30 | 34
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 23 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 13
White blood cell count decreased (Investigations) | 32 | 20
Neutrophil count decreased (Investigations) | 27 | 19
Weight decreased (Investigations) | 22 | 22
Platelet count decreased (Investigations) | 24 | 18
Blood alkaline phosphatase increased (Investigations) | 20 | 14
Lymphocyte count decreased (Investigations) | 23 | 9
Alanine aminotransferase increased (Investigations) | 8 | 15
Aspartate aminotransferase increased (Investigations) | 8 | 12
Headache (Nervous system disorders) | 32 | 31
Dizziness (Nervous system disorders) | 27 | 17
Dysgeusia (Nervous system disorders) | 17 | 17
Neuropathy peripheral (Nervous system disorders) | 22 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 | 5
Upper respiratory tract infection (Infections and infestations) | 15 | 6
Sepsis (Infections and infestations) | 12 | 7
Alpoecia (Skin and subcutaneous tissue disorders) | 50 | 19
Rash (Skin and subcutaneous tissue disorders) | 10 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 4
Palmer-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 12
Hypertension (Vascular disorders) | 6 | 30
Hypotension (Vascular disorders) | 16 | 13
Insomnia (Psychiatric disorders) | 17 | 17
Anxiety (Psychiatric disorders) | 14 | 11
Tachycardia (Cardiac disorders) | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT02049905/Prot_SAP_000.pdf